CLINICAL TRIAL: NCT02203370
Title: Cerebral Oximetry for Carotid EEA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Salzburger Landeskliniken (Other)
Responsible Party: Principal Investigator, Andreas Kokoefer, MD, Salzburger Landeskliniken
Other Study IDs: CerbralOximetry_01
Record Dates: First submitted 2014-07-24; First posted 2014-07-29 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2014-07

CONDITIONS: Carotid Thrombendarterectomy; Cerebral Oxygenation; NIRS; Regional Anesthesia
MeSH Terms: interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — S100B and NSE blood samples taken twice, before and after the surgical procedure
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- all patients: All patients will be measured throughout the procedure with both devices. There no further separation into groups as both sensors can be placed on the same patient.
  Interventions: Device: NIRS - Near-infrared spectroscopy

INTERVENTIONS:
Device: NIRS - Near-infrared spectroscopy
  Other Names: FORE-SIGHT™ Monitor (CAS Medical Systems, Branford, Connecticut, USA) and INVOS™ (Somanetics, Troy, Michigan, USA)

SUMMARY:
Aim oft he study is to compare two different devices for cerebral oximetry (FORE-SIGHTTM Monitor (CAS Medical Systems, Branford, Connecticut, USA and INVOSTM Somanetics, Troy, Michigan, USA) in patients undergoing surgical carotid thrombendarterectomy (cTEA) with crossclamped internal carotid artery (ACI). All procedures will be performed in regional anesthesia, therefore the patients will be awake and direct neurological examination during the procedure will be possible, giving information how the drop in cerebral saturation (measured with INVOS and FORESIGHT both on the same patient) correlates with any clinical symptoms.

We expect to see a difference in the total drop and in the delay of the drop of cerebral oxygen saturation, making it possible to detect varieties in specificity and sensitivity of both devices compared to neurologic examination in the awake patient.

ELIGIBILITY:
Inclusion Criteria:

- Patients with electively scheduled carotid thrombendarterectomy in regional anesthesia

Exclusion Criteria:

* refusing participation
* age <18 years
* pregnancy
* any contraindication to regional anesthesia or the use of NIRS
* participation in any other study affecting the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients scheduled for CTEA at the University Hospital Salzburg
Sampling Method: Non-Probability Sample
Enrollment: 126 (Estimated)
Dates: Start 2014-07; Primary Completion 2015-07 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
absolute tissue saturation (StO2) measured with(FORE-SIGHTTM Monitor (CAS Medical Systems, Branford, Connecticut, USA and INVOSTM Somanetics, Troy, Michigan, USA) | During the surgical procedure
  The drop in StO2 will be compared to the occurrence of any clinical i.e. neurological symptoms during clamping o the carotid artery while cTEA is performed.

SECONDARY OUTCOMES:
NSE | Before and after the surgery
  Biomarker for ischemic brain damage. Serum levels neuron specific enolase (NSE) increases in patients during the acute phase of brain damage. Therefore it is measured to find out whether or not there is correlation to a low oxygen saturation without neurological symptoms during cTEA.
S100B | Before and after the surgery
  Biomarker for ischemic brain damage. Serum levels of S100B increases in patients during the acute phase of brain damage. Therefore it is measured to find out whether or not there is correlation to a low oxygen saturation without neurological symptoms during cTEA.

OTHER OUTCOMES:
Hemodynamic parameters | During the surgical procedure
  Blood pressure
Hemodynamic parameters | During the surgical procedure
  Peripheral oxygen saturation
Hemodynamic parameters | During the surgical procedure
  ECG

CONTACTS AND LOCATIONS:
Overall Officials: Andreas Koköfer, M.D., Principal Investigator — UK für Anästhesiologie, LKH Salzburg
Locations (1):
- LKH University Clinic Salzburg, Salzburg, Salzburg, Austria